CLINICAL TRIAL: NCT01839084
Title: Impact of Xenon-anesthesia on the Renal Function After Partial Nephrectomy - PaNeX: Partial Nephrectomy Under Xenon:a Pilot Study
Brief Title: PaNeX: Partial Nephrectomy Under Xenon
Acronym: PaNeX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-051; 2012-005698-30 (EudraCT Number)
Record Dates: First submitted 2013-04-09; First posted 2013-04-24 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Renal Function After Partial Nephrectomy
Keywords: Xenon; Isoflurane; Anesthetics, Inhalation; Nephroprotection; Partial nephrectomy; Xenon versus Isoflurane anesthesia
MeSH Terms: conditions — Respiratory Aspiration | interventions — Xenon; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xenon (Experimental): Gaseous anesthetic, dosage: 60% (v/v) in 40% oxygen, continuous application during surgery
  Interventions: Drug: Xenon
- Isoflurane (Active Comparator): Inhalative anesthetic, dosage: 1.2% (v/v) in 40% oxygen/medical air , continuous application during surgery
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Xenon — general anaesthesia with xenon 60% in oxygen (FiO2=0.4)
  Other Names: Lenoxe
  Arms: Xenon
Drug: Isoflurane — general anesthesia with isoflurane 1.2% in 40% oxygen/medical air
  Other Names: Forene
  Arms: Isoflurane

SUMMARY:
Purpose of this study is to determine whether Xenon - as compared to Isoflurane - shows a nephroprotection after partial nephrectomy.

DETAILED DESCRIPTION:
A partial nephrectomy is accompanied by ischemia time, followed by reperfusion. This frequently leads to a kidney injury of the remained tissue and decrease of the renal function after surgery. As it was shown that Xenon has protective properties against ischemia/reperfusion injury, the investigators hypothesize that Xenon application during partial nephrectomy leads to a stronger nephroprotection than an anesthesia with Isoflurane.

The study will be conducted by two investigator types: The study enrollment and the post-anesthesia follow-up will be performed by Investigator I who is blinded to the study treatment. Investigator II will only perform general anesthesia for partial nephrectomy and will therefore necessarily be unblinded to the treatment conditions.

Patients will be randomly assigned to one of the following study groups. Group 1 (Xenon) will receive Xenon for maintenance of balanced anesthesia for partial nephrectomy. Group 2 (Isoflurane) will receive Isoflurane for the same surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and able to complete the requirements of this study
* Patients with renal carcinoma restricted to one kidney
* Patients undergoing partial nephrectomy
* Men and women >= 18 yrs
* Informed consent

Exclusion Criteria:

* Chronic renal failure with a GFR < 60ml/min/1,73m2 body surface area
* American Society of Anesthesiologists (ASA)>III
* Hypersensitivity to the study anaesthetics
* Chronic obstructive pulmonary disease (COPD) GOLD IV
* Acute coronary syndrome during the last 24 hours; haemodynamic instability, requirement of inotropic support
* Severe cardial dysfunction New York Heart Association (NYHA) >III
* Disabling neuropsychiatric disorders
* Increased intracranial pressure
* pregnant or breastfeeding women
* Women of childbearing potential
* Presumed uncooperativeness or legal incapacity
* Lack of informed consent
* Participation in a concomitant trial within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the impact of xenon-anesthesia on the renal function after partial nephrectomy, compared to an isoflurane-anesthesia. | Within the first 7 postoperative days
  Evaluation of the maximum decrease of glomerular filtration rate (GFR) within 7 days after partial nephrectomy surgery. Maximum decrease will be assessed by the difference between the baseline value of GFR and the minimum value of GFR after surgery.

SECONDARY OUTCOMES:
Secondary efficacy criteria for using xenon-anaesthesia during partial nephrectomy. | Intraoperatively
  Ischaemia time
Secondary efficacy criteria for using xenon-anaesthesia during partial nephrectomy. | Intraoperatively
  Duration of xenon/isoflurane exposition before and after the kidney ischemia time.
Secondary efficacy criteria for using xenon-anaesthesia during partial nephrectomy. | Intraoperatively until discharge from hospital
  Tumor size and histology, if applicable detection of hypoxia-inducible factor 1α (HIF-1α) in healthy resection border tissue
Secondary efficacy criteria for using xenon-anaesthesia during partial nephrectomy. | Intraoperatively and within the first 7 postoperative days
  Measurement of macrophage migration inhibitory factor (MIF) in serum
Secondary efficacy criteria for using xenon-anaesthesia during partial nephrectomy. | preaoperativ and Within the first 7 postoperative days
  Course of GFR determined with the Cystatin C value in serum
Secondary efficacy criteria for using xenon-anaesthesia during partial nephrectomy. | preaoperativ and Within the first 7 postoperative days
  Course of creatinine value in serum
Secondary efficacy criteria for using xenon-anaesthesia during partial nephrectomy. | Within the first 7 postoperative days
  Urine output within the first 48houres after surgery
Secondary efficacy criteria for using xenon-anaesthesia during partial nephrectomy. | Within the first 7 postoperative days
  If applicable determination of kidney injury molecule-1 (KIM-1)or neutrophil gelatinase-associated lipocalin (NGAL)
Secondary efficacy criteria for using xenon-anaesthesia during partial nephrectomy. | Within the first 7 postoperative days
  Determination of acute kidney failure according to the AKIN classification
Safety criteria for using xenon-anaesthesia during partial nephrectomy. | intraoperative
  Doses and concentration of study treatments
Safety criteria for using xenon-anaesthesia during partial nephrectomy. | intraoperative and within the first 7 postoperative days
  The peri-anaesthetic respiratory profile
Safety criteria for using xenon-anaesthesia during partial nephrectomy. | intraoperative and within the first 7 postoperative days
  The peri-anaesthetic haemodynamic profile
Safety criteria for using xenon-anaesthesia during partial nephrectomy. | intraoperative
  Intra-operative blood loss
Safety criteria for using xenon-anaesthesia during partial nephrectomy. | intraoperative and within the first 7 postoperative days
  The incidence of adverse event (AE) and serious adverse event (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Fahlenkamp, Dr. med., Principal Investigator — Department of Anesthesiology, University Hospital Aachen
Locations (1):
- Department of Anesthesiology, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Schafer P, Fahlenkamp A, Rossaint R, Coburn M, Kowark A. Better haemodynamic stability under xenon anaesthesia than under isoflurane anaesthesia during partial nephrectomy - a secondary analysis of a randomised controlled trial. BMC Anesthesiol. 2019 Jul 9;19(1):125. doi: 10.1186/s12871-019-0799-2. PMID 31288740
- [Derived] Stevanovic A, Schaefer P, Coburn M, Rossaint R, Stoppe C, Boor P, Pfister D, Heidenreich A, Christ H, Hellmich M, Fahlenkamp AV. Renal function following xenon anesthesia for partial nephrectomy-An explorative analysis of a randomized controlled study. PLoS One. 2017 Jul 18;12(7):e0181022. doi: 10.1371/journal.pone.0181022. eCollection 2017. PMID 28719609